CLINICAL TRIAL: NCT04764864
Title: Randomized Multicenter Study on the Management of Pelvic Fractures in Polytraumatized Patients With Hemodynamic Instability: Angioembolization vs Preperitoneal Packing
Brief Title: Pelvic Fractures in Polytraumatized Patients With Hemodynamic Instability: Angioembolization vs Preperitoneal Packing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No financing
Sponsor: Nuria Llorach-Perucho (Other)
Collaborators: Corporacion Parc Tauli (Other)
Responsible Party: Sponsor-Investigator, Nuria Llorach-Perucho, Principal Investigator, Corporacion Parc Tauli
Organization: Corporacion Parc Tauli (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PELVITRAU
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Trauma; Pelvic Fracture; Hemodynamic Instability
Keywords: Trauma; Pelvis Fracture; Hypovolemic Shock; Preperitoneal Pelvic Packing; Angioembolization; Hemodynamic Instability
MeSH Terms: conditions — Wounds and Injuries; Hip Fractures; Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angioembolization (Active Comparator)
  Interventions: Procedure: Angioembolization
- Preperitoneal Pelvic Packing (Active Comparator)
  Interventions: Procedure: Preperitoneal Pelvic Packing

INTERVENTIONS:
Procedure: Angioembolization — Via the femoral route, a non-selective pelvic arteriography with a selective embolization of the arterial branches that show direct or indirect signs of injury will be performed.
  In the event of persistent hemodynamic instability after selective embolization, non-selective bilateral embolization of the internal iliac arteries will be evaluated.
  The material used will vary depending on the characteristics of the injury and the availability of the materials.
  Arms: Angioembolization
Procedure: Preperitoneal Pelvic Packing — Pfannestiel incision / infraumbilical laparotomy. Dissection of tissues up to and including the transversalis fascia. Inferior to this and anterior to the peritoneum, the preperitoneal cavity is identified.
  Inclusion of radiopaque laparotomy gauze in each hemipelvis, from the posterior part (anterior to the sacro-iliac joint) to the most anterior in the retropubic position. Subsequently, the closure is carried out to increase the plugging effect.
  A second intervention is required to remove the material in 24-48 hours.
  Arms: Preperitoneal Pelvic Packing

SUMMARY:
Pelvic fracture is a usual injury in trauma patients. An unstable trauma patient with a pelvic fracture has an elevated risk of death due to pelvic bleeding and the associated injuries. Traditionally, it has been estimated that the main source of bleeding is venous and, consequently, the main treatment has been the preperitoneal pelvic packing. Nevertheless, according to new data, arterial bleeding appears to be a more important source of pelvic bleeding than it was thought and angioembolization seems to be a good alternative in the treatment of these injuries. Consequently, it is important to define better the management of these patients.

This investigation project consists in a clinical trial study, performed by a multidisciplinary team of many hospitals around the country, in which angioembolization and preperitoneal pelvic packing are compared. Unstable trauma patients with a pelvic fracture and no other injuries (negative FAST / peritoneal aspiration, no evidence of bone fractures or thoracic injuries) will be submitted, in less than 60 minutes from hospital arrival, to angioembolization or preperitoneal pelvic packing, according to randomization. There will be a specific timing evaluation of different markers: hemodynamic (vital signs at arrival, immediately and 24 hours after treatment) and analytic (at arrival and upon entering to the Intensive Care Unit). Registered variables include: blood cell transfusions, vasoactive drug requirements, time elapsed between hospital admission and intervention, treatment duration, need of other strategies to stop pelvic bleeding, complications and mortality.

The objective of this study is to determinate if angioembolization is superior to preperitoneal pelvic packing for pelvic bleeding control in unstable trauma patients due to pelvic bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure ≤ 90 mmHg
* Heart rate > 100 bpm
* Shock Index ≥ 0,8
* Pelvic fracture
* Negative FAST / peritoneal aspiration

Exclusion Criteria:

* Other causes of bleeding that require treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Pelvic bleeding control based on clinical response | 24 hours
  Clinical response after the intervention

SECONDARY OUTCOMES:
Additional techniques | Through study completion, an average of 2 years
  Need for additional techniques after the intervention to control bleeding associated with pelvic fracture
Post-procedure complications | Through study completion, an average of 2 years
  Presence of post-procedure complications
Post-procedure complications degree | Through study completion, an average of 2 years
  Description of post-procedure complications: Clavien Dindo scale
Post-procedure complications degree | Through study completion, an average of 2 years
  Description of post-procedure complications: Comprehensive Complication Index
Mortality | Through study completion, an average of 2 years
  Death of the pacient (cause and date)
Blood cell transfusion | Through study completion, an average of 2 years
  Need for blood cell transfusion for patients (number and need for masive transfusion protocol activation)
Time until intervention | Time until intervention (up to 60 minutes)
  Time elapsed between hospital admission and intervention

OTHER OUTCOMES:
Time until arrival at hospital | Time until arrival at hospital (up to 30 minutes)
  Time elapsed between prehospital attention and hospital admission
Duration of angioembolization | Through study completion, an average of 2 years
  Duration of angioembolization
Angioembolization treatment | Through study completion, an average of 2 years
  Arteries treated with angioembolization
Duration of Preperitoneal Pelvic Packing | Through study completion, an average of 2 years
  Duration of Preperitoneal Pelvic Packing
Intensive care unit stay | Through study completion, an average of 2 years
  Number of days that the patient remains in the intensive care unit
Hospital stay | Through study completion, an average of 2 years
  Number of days that the patient remains in hospital
Readmission | 30 days after discharge
  Readmission 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Llorach-Perucho, MD, Principal Investigator — Corporacion Parc Tauli; Salvador Navarro-Soto, MD, PhD, Study Director — Corporacion Parc Tauli; Andrea Campos-Serra, MD, Study Director — Corporacion Parc Tauli
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain